CLINICAL TRIAL: NCT00859430
Title: A Single-Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalence Study of Levetiracetam 1000 mg Tablet Under Fed Conditions
Brief Title: Levetiracetam 1000 mg Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-117-SA
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Experimental): Levetiracetam 1000 mg Tablet (test) dosed in first period followed by Keppra® 1000 mg Tablet (reference) dosed in second period
  Interventions: Drug: Levetiracetam
- Keppra® (Active Comparator): Keppra® 1000 mg Tablet (reference) dosed in first period followed by Levetiracetam 1000 mg Tablet (test) dosed in second period
  Interventions: Drug: Keppra®

INTERVENTIONS:
Drug: Levetiracetam — 1000 mg Tablet
  Arms: Levetiracetam
Drug: Keppra® — 1000 mg Tablet
  Arms: Keppra®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of an investigational formulation of levetiracetam 1000 mg tablet to an equivalent oral dose of the commercially available reference product under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

All subjects must satisfy the following criteria to be considered for study participation:

* Subject must be male or non-pregnant, non-breast-feeding female
* Subject must be at least 18 years of age
* Subject must have a Body Mass Index (BMI) between 19 and 30 kg/m2, inclusive, and body weight should be at least 50 kg (110 lbs)
* Female Subjects - not surgically sterile or at least two years postmenopausal - must agree to utilize one of the following forms of contraception, if sexually active with a male partner, from screening through completion of the study. Approved forms of contraception are abstinence, double barrier (condom with spermicide, diaphragm with spermicide), intra-uterine device (IUD), or vasectomized partner (6 months minimum since vasectomy).
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to the start of any study-specific procedures.
* Subject is willing and able to consume the entire high-calorie, high-fat breakfast meal in the designated timeframe required during each study period.
* Subject is willing and able to remain in the study unit for the entire duration of each confinement period and return for any outpatient visits.

Exclusion Criteria

Subjects may be excluded for any of the following:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition which, in the opinion of the Investigator would jeopardize the safety of the subject or the validity of the study results.
* Has a clinically significant abnormal finding on the physical exam, medical history, ECG or clinical laboratory results at screening.
* History or presence of allergic or adverse response to levetiracetam or related drugs.
* Has been on a significantly abnormal diet during the four weeks preceding the first dose of study medication.
* Has donated blood or plasma within 30 days prior to the first dose of study medication.
* Has participated in another clinical trial within 30 days prior to the first dose of study medication.
* Has used any over-the-counter (OTC) medication, including nutritional supplements, within 7 days prior to the first dose of study medication.
* Has used any prescription medication, including hormonal contraceptive or hormonal replacement therapy, within 14 days prior to the first dose of study medication.
* Has been treated with any known enzyme altering drugs such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication.
* Has smoked or used tobacco products within 90 days prior to the first dose of study medication.
* Subject has consumed alcohol, caffeine/xanthine, or grapefruit containing beverages and foods from 48 hours prior to the dose of study medication and throughout the sample collection period.
* Is a female with a positive pregnancy test result.
* Female who has used implanted or injected hormonal contraceptives anytime during the 6 months prior to study start.
* Has an intolerance to venipuncture.
* Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates)
* Has a history of drug or alcohol abuse.
* Has had a positive test for, or has been treated for hepatitis B, hepatitis C or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P Doherty, D.O., Principal Investigator — CEDRA
Locations (1):
- CEDRA Clinical Research, LLC, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Levetiracetam (Test) First: Levetiracetam 1000 mg Tablet (test) dosed in first period followed by Keppra® 1000 mg Tablet (reference) dosed in second period
- Keppra® (Reference) First: Keppra® 1000 mg Tablet (reference) dosed in first period followed by Levetiracetam 1000 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Levetiracetam (Test) First | Keppra® (Reference) First
Started | 11 | 11
Completed | 11 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Levetiracetam (Test) First | Keppra® (Reference) First
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam (Test) First | Keppra® (Reference) First | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 6 | 9 | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 8 | 10 | 18
  Black | 1 | 0 | 1
  American Indian or Alaska Native | 1 | 1 | 2
  Multi-Racial | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Levetiracetam: Levetiracetam 1000 mg Tablet (test) dosed in either period
- Keppra®: Keppra® 1000 mg Tablet (reference) dosed in either period
Arm/Group | Levetiracetam | Keppra®
Number analyzed (Participants) | 21 | 21
mcg/mL | 26.320 (5.060) | 24.927 (4.427)
Statistical Analysis 1: Comparison: Levetiracetam vs Keppra®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Ratio of Geometric Means = 105, 90% CI [98.6 to 112] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Levetiracetam | Keppra®
Number analyzed (Participants) | 21 | 21
mcg*h/mL | 261.018 (45.320) | 263.968 (40.007)
Statistical Analysis 1: Comparison: Levetiracetam vs Keppra®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Ratio of Geometric Means = 98.6, 90% CI [96.2 to 101] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 36 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Levetiracetam | Keppra®
Number analyzed (Participants) | 21 | 21
mcg*h/mL | 249.260 (44.183) | 252.523 (39.858)
Statistical Analysis 1: Comparison: Levetiracetam vs Keppra®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Ratio of Geometric Means = 98.4, 90% CI [95.9 to 101] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.